CLINICAL TRIAL: NCT05478070
Title: The Use of Continuous Glucose Monitors in the Care of Pregnant and Postpartum Women to Limit Frequency of Staff Exposure and Preserve Staff Personal Protective Equipment
Brief Title: Continuous Glucose Monitoring for Personal Protective Equipment Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ohio State University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020H0182
Record Dates: First submitted 2022-04-21; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus (DM)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Dexcom CGM (Other): Proof of concept randomized study to evaluate the utility of Dexcom-G6 continuous glucose monitors for assessment of glycemic control in pregnant and postpartum women with insulin-requiring diabetes mellitus during hospitalizations
  Interventions: Device: Dexcom G6

INTERVENTIONS:
Device: Dexcom G6 — Continuous glucose monitor

SUMMARY:
Diabetes mellitus (DM) affects roughly 8% of pregnancies and is associated with significant perinatal and maternal morbidity. Current obstetric practice is complicated by the emergence of the SARS-COV-2 pandemic, resulting in morbidity and mortality secondary to complications of COVID-19. Care coordination among the teams caring for women admitted for antepartum, intrapartum, and postpartum care with suspected or confirmed COVID-19 is required to conserve PPE and minimize staff exposure. The investigators propose a pilot proof of concept randomized study to evaluate the utility of Dexcom-G6 continuous glucose monitors for assessment of glycemic control in pregnant and postpartum women with insulin-requiring diabetes mellitus during hospitalizations, as a proof of concept in the efforts to reduce the number of point of care glucose tests needed, reduce staff exposure, and conserve PPE use.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-50 years with a viable singleton or twin intrauterine pregnancy between 8 0/7 and 41 6/7 weeks gestation based on the best obstetric estimate by ACOG criteria
* Diagnosis of pre-gestational or gestational diabetes mellitus A2, admitted to the hospital for labor or other antepartum admissions (besides DKA or glucoregulation)
* Able to understand the study, and having understood, provide written informed consent in English
* Infants who survive to hospital discharge who are born to women enrolled in the study

Exclusion Criteria:

* Participation in another trial that may influence the primary outcome, without prior approval
* Higher order pregnancy
* History of severe skin allergy to adhesive products or CGM
* DKA, admission for glucoregulation
* COVID-19 PUI or confirmed positive

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Maternal outcomes | 1 year
  Outcomes pertaining to overall maternal health based on glucose control as determined by HbA1c
Neonatal outcomes | 1 year
  Outcomes pertaining to overall neonatal health based on incidence of neonatal diseases upon birth as determined by a physical exam of the neonate
Maternal outcomes | 1 year
  Outcomes pertaining to overall maternal health based on glucose control as determined by serum glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Buschur, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No